CLINICAL TRIAL: NCT03546543
Title: The Effects of Prone Versus Supine Position on the Oxygenation Instability of Premature Infants as Documented by SpO2 Histograms
Brief Title: The Effects of Position on the Oxygenation Instability of Premature Infants as Documented by SpO2 Histograms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Liron Borenstein MD, Doctor, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 0167-17-RMB
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Premature Infant; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine (Experimental)
  Interventions: Procedure: Position change
- Prone (Experimental)
  Interventions: Procedure: Position change

INTERVENTIONS:
Procedure: Position change — Each subject will serve as his or her own control. Half of the infants will be placed supine for 3 hours, followed by 3 hours of prone positioning and back to supine for 3 hours and the other half will be start in prone position with consecutive periods of supine and then prone

SUMMARY:
SpO2 instability is in the nature of premature infants. Hypoxic episodes occur spontaneously in many of these infants, especially after the first week of life. Different interventions have been shown to influence the incidence of hypoxemic episodes in premature infants. A few studies point towards potential clinical benefits of better oxygenation and less hypoxic events by positioning very low birth weight infants prone, though a recent meta-analysis didn't find a clear benefit of prone position.

The aim of this study is to evaluate the changes in oxygenation among preterm infants receiving respiratory support when positioned prone versus supine, as documented by SpO2 histograms.

ELIGIBILITY:
Inclusion Criteria:

Premature infants with a weight < 1500 g who are receiving respiratory support

Exclusion Criteria:

Congenital anomalies, acute lung pathology for example x-ray confirmed pneumonia, air leak, active culture proven sepsis or on inotropic support for low blood pressure.

Min Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation instability | 3 hours in each position
  SPO2 histogram documents the oxygenation stability. we will record the histogram at the end of each period of time and compare it

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No